CLINICAL TRIAL: NCT04087278
Title: Cardiovascular Health Arterial Stiffness Raspberry and Microbiome (CHARM)
Acronym: CHARM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Centro de Edafología y Biología Aplicada del Segura (Other Government); Washington Red Raspberry Commission (Other)
Responsible Party: Principal Investigator, Dr Ana Rodriguez-Mateos, Reader in Nutritional Sciences, King's College London
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CHARM Study
Record Dates: First submitted 2019-09-02; First posted 2019-09-12 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers
Keywords: Cardiovascular system; Polyphenols

STUDY DESIGN:
Intervention Model Description: Double-blind placebo randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Metabotype A (Active Comparator): Taking treatment
  Interventions: Dietary Supplement: Red Raspberry Ellagitannin Extract
- Metabotype B (Active Comparator): Taking treatment
  Interventions: Dietary Supplement: Red Raspberry Ellagitannin Extract
- Metabotype 0 (Active Comparator): Taking treatment
  Interventions: Dietary Supplement: Red Raspberry Ellagitannin Extract
- Placebo (Placebo Comparator): Taking matching placebo
  Interventions: Dietary Supplement: Matching Placebo

INTERVENTIONS:
Dietary Supplement: Red Raspberry Ellagitannin Extract — Purified red raspberries ellagitannins extract 560 mg (4 capsules/day)
  Arms: Metabotype 0; Metabotype A; Metabotype B
Dietary Supplement: Matching Placebo — Placebo treatment matching intervention (no ellagitannin) 560 mg (4 capsules/day)
  Arms: Placebo

SUMMARY:
In this study, the investigators aim to determine the health benefits of red raspberry ellagitannin consumption on cardiovascular health. The study population is stratified according to the urolithin metabotypes (gut-microbial metabolic profile): UM-0, UM-A and UM-B.

The investigators will evaluate changes in blood pressure, endothelial function, arterial stiffness, lipid profile, cognitive performance and gut microbiome composition.

DETAILED DESCRIPTION:
Red raspberries are a good source of polyphenols including ellagitannins. Previous work suggests that urolithins, gut microbial metabolites derived from ellagitannins contained in raspberries, can improve vascular health. It has also been observed that the capacity of the gut microbiome to metabolize urolithins can influence the cardiometabolic response to ellagitannin consumption. In this work the investigators aim to investigate whether urolithin metabotypes (UM-A, B and 0) can influence the vascular response to a (poly)phenol-rich breakfast containing red raspberry ellagitannins in a healthy UK population.

You will be stratified by metabotype in a first phase (NCT03573414) and are then randomly allocated to treatment or placebo. Outcomes are measured at baseline and after 12 weeks consumption of the study product.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women aged 20-70 years old
* BMI between 18.5-35 kg/m²
* Normotensive: SBP lower than 140 mmHg or DBP lower than 90 mmHg
* Willing to maintain their normal eating/drinking habits and exercise habits to avoid changes in body weight over the duration of the study
* Able to understand the nature of the study
* Able to give signed written informed consent

Exclusion Criteria:

* Have required treatment for hypertension at any time (e.g. statins, aspirin, blood pressure lowering drugs)
* BMI outside range
* Manifest cardiovascular disease including coronary artery disease, cerebrovascular disease and peripheral artery disease
* Currently treated with a diet
* Chronic-acute disease
* Unstable psychological condition
* Diabetes mellitus, metabolic syndrome, acute inflammation, terminal renal failure, malignancies or abnormal heart rhythm (lower or higher than 60-100 bpm)
* History of cancer, myocardial infarction, cerebrovascular incident or kidney abnormality
* Allergies to berries, flax seeds and soy milk or other significant food allergy
* Requiring chronic antimicrobial or antiviral treatment
* Reported having taken food supplements, dietary supplement or herbal remedies within 1 month of study start
* Weight loss of more than 10% body weight in the previous 6 months
* Reported participant in another study within one month before the study start
* Smoke an irregular amount of cigarettes per day or planning to quit smoking in the next 3 months
* Unable to tolerate breakfast ingestion
* Pregnant woman/ lactating woman/ woman planning to become pregnant/ premenopausal women who do not have a regular menstrual cycle/ premenopausal women who do not have adequate method of contraception
* Any reason or condition that in the judgment of the clinical investigator(s) may put the subject at unacceptable risk or that may preclude the subject from understanding or complying with the study's requirements
* Unable to swallow the capsule.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Change in flow-mediated dilation (FMD) | Baseline vs 12 weeks post-consumption
  Determine the effect of the Red raspberry ellagitannin extract vs Placebo on flow-mediated dilation at 12 weeks post consumption

SECONDARY OUTCOMES:
Change in office blood pressure | Baseline vs 12 weeks post-consumption
  Determine the effect of the Red raspberry ellagitannin extract vs Placebo on office systolic and diastolic blood pressure, at 12 weeks post consumption
Change in heart rate | Baseline vs 12 weeks post-consumption
  Determine the effect of the Red raspberry ellagitannin extract vs Placebo on heart rate, at 12 weeks post consumption
Change in blood flow velocity | Baseline vs 12 weeks post-consumption
  Determine the effect of the Red raspberry ellagitannin extract vs Placebo on blood flow velocity at 12 weeks post consumption
Change in pulse wave velocity (PWV) | Baseline vs 12 weeks post-consumption
  Determine the effect of the Red raspberry ellagitannin extract vs Placebo on pulse wave velocity (PWV) using a Sphygmocor device, at 12 weeks post consumption
Change in augmentation Index (AIx) | Baseline vs 12 weeks post-consumption
  Determine the effect of the Red raspberry ellagitannin extract vs Placebo on augmentation Index (AIx) using a Sphygmocor device, at 12 weeks post consumption
Change in blood lipid concentrations | Baseline vs 12 weeks post-consumption
  Determine the effect of the Red raspberry ellagitannin extract vs Placebo on blood lipids (Total, HDL and LDL cholesterol, triglycerides), at 12 weeks post consumption
Change in blood inflammatory markers (circulating concentrations) | Baseline vs 12 weeks post-consumption
  Determine the effect of the Red raspberry ellagitannin extract vs Placebo on blood inflammatory markers (CRP, IL-6), at 12 weeks post consumption
Change in 24-hour heart rate | Baseline vs 12 weeks post-consumption
  Determine the effect of the Red raspberry ellagitannin extract vs Placebo on 24-hour heart rate, using a monitor, at 12 weeks post consumption
Change in 24-hour ambulatory blood pressure | Baseline vs 12 weeks post-consumption
  Determine the effect of the Red raspberry ellagitannin extract vs Placebo on 24-hour ambulatory blood pressure (SBP and DBP), using a monitor, at 12 weeks post consumption
Change in 24-hour AIx and PWV | Baseline vs 12 weeks post-consumption
  Determine the effect of the Red raspberry ellagitannin extract vs Placebo on 24-hour arterial stiffness (AIx and PWV), using a monitor, at 12 weeks post consumption

OTHER OUTCOMES:
Change in urinary metabolic (poly)phenol metabolite concentrations | Baseline vs 12 weeks post-consumption
  Measured by liquid chromotography-mass spectrometry (LC/MS) at baseline and after 12 weeks in a 24h urine sample
Change in plasmatic metabolic (poly)phenol metabolite concentrations | Baseline vs 12 weeks post-consumption
  Measured by liquid chromotography-mass spectrometry (LC/MS) at baseline and after 12 weeks
Gut microbiome composition | Baseline vs 12 weeks post-consumption
  Analysis of the microbiome composition and diversity at baseline and after 12 weeks post-consumption
Change in verbal-episodic memory performance assessed by AVLT | Baseline vs 12 weeks post-consumption
  Assessment of the performance with the difference of words remembered between baseline and after 12 weeks post-consumption.
Change in executive function performance assessed by the switching task | Baseline vs 12 weeks post-consumption
  Assessment of the performance calculating the difference in mistakes (not applying the right rule when needed) between baseline and after 12 weeks post-consumption.
Change in visual-spatial working memory performance assessed by the Corsi task | Baseline vs 12 weeks post-consumption
  Assessment of the performance with the difference in mistakes remembering the block patterns between baseline and after 12 weeks post-consumption.
Change in mood using the PANAS questionnaire | Baseline vs 12 weeks post-consumption
  Assessment of the change in the mood using the PANAS questionnaire containing 10 positive affects and 10 negative affects rated using a 5-point likert scale that ranges from "(1) Not at all to (5) Extremely", between baseline and after 12 weeks post-consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Rodriguez-Mateos, PhD, Principal Investigator — King's College London
Locations (1):
- Department of Nutritional Sciences, School of Life Course Sciences, Faculty of Life Sciences and Medicine, King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No